CLINICAL TRIAL: NCT07160790
Title: Efficacy and Safety of JP-1366 in Patients With Non-erosive Gastroesophageal Reflux(NERD) Disease: Double-blind, Randomized
Brief Title: Phase 3 Study of JP-1366: Efficacy and Safety of JP-1366 in Patients With Non-erosive Gastroesophageal Reflux Disease
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Onconic Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JP-1366-305
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Non-erosive Gastroesophageal Reflux Disease
Keywords: Non-erosive Reflux Disease; Non-Erosive Gastro-Esophageal Reflux Disease
MeSH Terms: conditions — Non-Erosive Reflux Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: JP-1366 A mg + Placebo (Experimental)
  Interventions: Drug: JP-1366 + placebo
- Group 2: JP-1366 B mg + Placebo (Experimental)
  Interventions: Drug: JP-1366 + placebo
- Placebo + Placebo (Placebo Comparator)
  Interventions: Drug: Placebo + Placebo

INTERVENTIONS:
Drug: JP-1366 + placebo — taking JP-1366 + placebo
  Arms: Group 1: JP-1366 A mg + Placebo; Group 2: JP-1366 B mg + Placebo
Drug: Placebo + Placebo — taking placebo + placebo
  Arms: Placebo + Placebo

SUMMARY:
This study aims to evaluate the efficacy and safety of JP-1366 in Patients with NERD

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have experienced both heartburn and acid regurgitation
* Subjects in whom no mucosal breaks were observed on upper GI endoscopy at Visit 1 by LA Classification
* Subjects who fully understand this clinical trial and voluntarily signed the informed consent form

Exclusion Criteria:

* Subjects who have significant gastrointestinal diseases or procedures affecting the esophagus, stomach, or duodenum
* Subjects who have a history of recent substance abuse, malignancy, systemic autoimmune or immune deficiency diseases, refractory response to PPI/P-CAB, hypersensitivity to study drugs, genetic metabolic disorders, or significant psychiatric conditions.
* Subjects who showed clinically significant abnormalities in laboratory tests
* Positive result in the H. pylori test
* Pregnant or breast-feeding women
* Subjects who require hospitalization are scheduled to undergo surgery during the study period, or have undergone major surgery requiring general anesthesia
* Other people deemed unsuitable for participation in this study according to the medical opinion of the investigator

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 321 (Estimated)
Dates: Start 2025-09-02 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of days with no heartburn | The proportion of days with no heartburn for 24 hours (daytime/nighttime) over 4 weeks

IPD SHARING:
Plan to Share IPD: No